CLINICAL TRIAL: NCT01444833
Title: Molecular - Genetic Alterations in Adipose Tissue After Change in Therapy From ACE Inhibitors to AT1 Receptor Blockers in Patients With Essential Hypertension
Brief Title: Changes After Angiotensin Converting Enzyme (ACE) Inhibitor Replacement by Angiotensin II Receptor Type I (AT1) Blocker
Acronym: ADIRAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Stefan Zorad, Head of Laboratory, Slovak Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MinHealth; 2007/27-SAV-02 (Other Grant/Funding Number: Slovak Ministry of Health)
Record Dates: First submitted 2011-09-19; First posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: hypertension; obesity; metabolism; angiotensin
MeSH Terms: conditions — Hypertension; Obesity | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Candesartan — 32 mg per day duration 6 months
  Other Names: Atacand

SUMMARY:
It is supposed that the significant metabolic effects (improvement of insulin sensitivity) of hypertension therapy with renin-angiotensin system (RAS) blockers in humans are mediated mainly via changes in abdominal adipose tissue. This project is aimed to confirm the hypothesis that increased concentrations of circulatory angiotensin II after angiotensin II receptor type I (AT1) blockade leads, via stimulation of angiotensin II receptor type II (AT2), to activation of adipogenesis and improvement of insulin sensitivity. Therefore, in hypertensive patients, the components of RAS and the parameters of insulin sensitivity on systemic (in plasma) and local (in adipose tissue and in its interstitial fluid) level will be studied. The main aim of the study is to identify the changes occurring in patient before and 6 months after the conversion of therapy from angiotensin converting enzyme (ACE) inhibitors to AT1 receptor blockers. Observed parameters will include gene expression of RAS components, parameters of insulin sensitivity, amount, and cellularity of adipose tissue obtained by biopsy, evaluation of direct production of cytokines and angiotensins into the interstitial fluid of fat tissue obtained by microdialysis and evaluation of the selected parameters in plasma.

DETAILED DESCRIPTION:
Arterial hypertension is nowadays considered a metabolic disease, due to its occurrence together with other risk factors of atherosclerosis like obesity, dyslipidemia, insulin resistance, impaired glucose regulation to diabetes mellitus type 2. These factors often result into the metabolic syndrome. Its pathogenetic mechanisms are not completely clarified yet, polygenic inheritance and environmental factors are probably involved. Therefore, from pathophysiological perspective of hypertension therapy a complex approach to the patient is needed. This approach requires the understanding of all known risk factors leading to the pharmacological and non-pharmacological intervention aimed to eliminate the risk factors of atherosclerosis. One of the main homeostatic systems participating in blood pressure regulation is the RAS.

The present pharmacotherapy provides the possibility to influence the RAS through the inhibition of a) renin, b)ACE or c) through blockade of AT1 receptors.

1. Renin inhibitors belong to the recent therapeutic approaches in hypertension treatment. Clinical studies, which could enable their use in daily practice, have not been completed yet.
2. Inhibition of angiotensin converting enzyme prevents the transformation of angiotensin I (Ang I) to angiotensin II (Ang II), prevents the breakdown of vasodilatatory kinins, mainly bradykinin, leading to the NO-mediated vasodilatation. The positive effects of therapy with ACE inhibitors are based besides the decrease of circulating Ang II also on decreased influence of tissue Ang II, mainly in the vascular wall and on diminished norepinephrine release from neural terminals of autonomic nervous system (Noshiro et al. 1991). The ACE inhibitors reduce plasma Ang II levels, thus the AT1 and AT2 receptors are less stimulated by the hormone leading to upregulation of the homologue ACE2, thereby increasing the production of angiotensin (1-7) (Ferrario et al. 2005). Angiotensin (1-7) binds to the AT1 as well as to the AT2 receptors and to its tentative AT(1-7) receptor.

   Some ACE inhibitors have a positive effect on improvement of glucose metabolism. The mechanism of improvement of insulin sensitivity has not been completely explained yet. It is supposed, that the positive insulin-sensitizing effects of ACE inhibitors could be mediated by hemodynamic changes - by improvement of skeletal muscle blood flow and/or by stimulation of insulin signaling pathways or by increasing the expression and the number of glucose transporter GLUT4. The improvement of insulin sensitivity during the therapy with ACE inhibitors correlated with the changes in the ion calcium/magnesium balance. The sympatholytic effect of the therapy with RAS inhibitors could also positively influence the metabolic parameters, supported by a study showing a decrease in serum epinephrine and an increase of insulin stimulated glucose uptake in normotensive volunteers treated with ACE inhibitor. In animal models of hypertension, the ACE inhibitors had a positive effect on reduction of free fatty acids levels and therefore a positive effect on insulin action.
3. AT1 receptor blockade (by sartans) results in elevated plasma Ang II concentrations and to preferential stimulation of AT2 receptors. Compared to AT1, stimulation of AT2 receptors exerts an antagonistic effect by inducing vasodilatation, apoptosis, and by inhibiting growth and proliferation of vascular smooth muscle cells. In addition, high Ang II concentrations seem to upregulate low levels or even re-express missing AT2 receptors in adult rat adipose tissue. ACE2 expression is also upregulated under AT1 blockade thus increased concentrations of angiotensin (1-7) in vivo in humans are assumed even not studied yet. Angiotensin (1-7) binds preferentially to non-blocked AT2 receptors evoking additional depressor activity via kinin/NO/cGMP cascade inducing vasodilatation and improvement in hemodynamics.

Overall, ACE inhibition exerts its beneficial effects on blood pressure via decreased Ang II concentrations and elevated bradykinin. On the other hand, blockade of AT1 receptors causes simultaneous overstimulation of AT2 receptors by elevated concentrations of Ang II, angiotensin (1-7) and angiotensin A having a positive effect on adipogenesis resulting in changes of regulatory mechanisms influencing the insulin action.

The sartans have an insulin-sensitizing effect; their exact mechanism is unknown so far. Some of the AT1 receptor blockers display a weak peroxisome proliferator activator receptor (PPARγ) agonist activity which might promote the adipocyte differentiation. However, sartans without the PPARγ-agonist activity have a significant effect on adipocyte downsizing and improvement of insulin sensitivity markers as well. These results suggest that there may be a distinct mechanism, other than direct activation of PPARγ that is responsible for adipocyte differentiation and improvement of metabolic parameters.

It is supposed that adipose tissue, except from systemic hemodynamic and sympatholytic effect is responsible for the insulin-sensitizing effect of sartans. In the last 20 years, the adipose tissue has been well studied, since it is no more considered only an energy storage but also a source of several substances - hormones, enzymes and bioactive peptides generally called adipokines.

Human and rat adipose tissue contains complete local renin-angiotensin system (RAS). Components of adipose RAS undergo significant changes when the amount of adipose tissue and the adipocyte size enlarge. This leads to the assumption, that RAS plays an important role in regulation of adipose tissue mass. In vitro studies showed that Ang II inhibits adipocyte differentiation resulting in increased proportion of large insulin-resistant adipocytes and ectopic lipid deposition in other tissues. In the large adipocytes, expression and production of TNF is increased and adiponectin secretion inhibited through AT1 receptors. TNF is a cytokine impairing insulin action, highly expressed in adipose tissue in obesity and metabolic syndrome. It is known that the insulin sensitivity of adipocytes decreases with their size. RAS blockade stimulates adipogenesis in adipose tissue, probably via stimulation of AT2 receptors resulting in increased number of small insulin-sensitive cells. Several authors have observed a decrease in adipocyte size in retroperitoneal and epididymal adipose tissue in line with improved insulin sensitivity after RAS blockade in rats. Blockade of AT1 receptors in co-culture of human preadipocytes and adipocytes leaded also to increased adipogenesis. It is assumed that in vivo blockade of RAS might result in increased proportion of small adipocytes due to adipogenesis with simultaneous decrease in number of large cells due to apoptosis. The increased proportion of smaller adipocytes is reflected in changes of expression and release of adipokines producing more adiponectin and less TNF. Indeed, blockade of RAS elevates serum concentrations of adiponectin in patients with essential hypertension. In rats, serum concentrations as well as mRNA expression of adiponectin and PPARγ in adipose tissue increased. PPARγ plays probably a role in mechanisms related to the effect of RAS inhibition on changes in adipose tissue amount and its insulin sensitivity. In vivo in human body, to our knowledge these changes in production of RAS components in relation to adiposity and cellularity of the adipose tissue, to adipokines secretion and to parameters of insulin sensitivity have not been studied yet.

ELIGIBILITY:
Inclusion Criteria:

* essential hypertension
* ACE inhibitors

Exclusion Criteria:

* diabetes mellitus
* endocrinopathies
* no smokers

Ages: 25 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Systemic Insulin Sensitivity after Replacement of ACE Inhibitor by AT1 Blocker | 6 months
  Oral glucose tolerance test (OGTT) will be used to determine systemic insulin sensitivity.

SECONDARY OUTCOMES:
Adipocyte Diameter from Subcutaneous Adipose Tissue after Replacement ACE Inhibitor by AT1 Blocker | 6 months
  The tissue obtai ned by biopsy will be digested by collagenase and the diameter of isolated adipocytes will be evaulated by light microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zorad, Dr., Principal Investigator — Institute of Experimental Endocrinology SAS
Locations (1):
- Institute of Experimental Endocrinology, SAS, Bratislava, Slovakia

REFERENCES:
- [Background] Zorad S, Dou JT, Benicky J, Hutanu D, Tybitanclova K, Zhou J, Saavedra JM. Long-term angiotensin II AT1 receptor inhibition produces adipose tissue hypotrophy accompanied by increased expression of adiponectin and PPARgamma. Eur J Pharmacol. 2006 Dec 15;552(1-3):112-22. doi: 10.1016/j.ejphar.2006.08.062. Epub 2006 Sep 9. PMID 17064684
- [Background] Santos RA, Simoes e Silva AC, Maric C, Silva DM, Machado RP, de Buhr I, Heringer-Walther S, Pinheiro SV, Lopes MT, Bader M, Mendes EP, Lemos VS, Campagnole-Santos MJ, Schultheiss HP, Speth R, Walther T. Angiotensin-(1-7) is an endogenous ligand for the G protein-coupled receptor Mas. Proc Natl Acad Sci U S A. 2003 Jul 8;100(14):8258-63. doi: 10.1073/pnas.1432869100. Epub 2003 Jun 26. PMID 12829792
- [Background] Scheen AJ. Renin-angiotensin system inhibition prevents type 2 diabetes mellitus. Part 2. Overview of physiological and biochemical mechanisms. Diabetes Metab. 2004 Dec;30(6):498-505. doi: 10.1016/s1262-3636(07)70147-7. PMID 15671919
- [Background] Sharma AM, Janke J, Gorzelniak K, Engeli S, Luft FC. Angiotensin blockade prevents type 2 diabetes by formation of fat cells. Hypertension. 2002 Nov;40(5):609-11. doi: 10.1161/01.hyp.0000036448.44066.53. PMID 12411451
- [Background] Walters PE, Gaspari TA, Widdop RE. Angiotensin-(1-7) acts as a vasodepressor agent via angiotensin II type 2 receptors in conscious rats. Hypertension. 2005 May;45(5):960-6. doi: 10.1161/01.HYP.0000160325.59323.b8. Epub 2005 Mar 14. PMID 15767466
- [Background] Weyer C, Foley JE, Bogardus C, Tataranni PA, Pratley RE. Enlarged subcutaneous abdominal adipocyte size, but not obesity itself, predicts type II diabetes independent of insulin resistance. Diabetologia. 2000 Dec;43(12):1498-506. doi: 10.1007/s001250051560. PMID 11151758
- [Background] Yamauchi T, Kamon J, Waki H, Murakami K, Motojima K, Komeda K, Ide T, Kubota N, Terauchi Y, Tobe K, Miki H, Tsuchida A, Akanuma Y, Nagai R, Kimura S, Kadowaki T. The mechanisms by which both heterozygous peroxisome proliferator-activated receptor gamma (PPARgamma) deficiency and PPARgamma agonist improve insulin resistance. J Biol Chem. 2001 Nov 2;276(44):41245-54. doi: 10.1074/jbc.M103241200. Epub 2001 Aug 31. PMID 11533050
- [Background] Yang X, Jansson PA, Nagaev I, Jack MM, Carvalho E, Sunnerhagen KS, Cam MC, Cushman SW, Smith U. Evidence of impaired adipogenesis in insulin resistance. Biochem Biophys Res Commun. 2004 May 14;317(4):1045-51. doi: 10.1016/j.bbrc.2004.03.152. PMID 15094374
- [Background] Zorad S, Fickova M, Zelezna B, Macho L, Kral JG. The role of angiotensin II and its receptors in regulation of adipose tissue metabolism and cellularity. Gen Physiol Biophys. 1995 Oct;14(5):383-91. PMID 8786038
- [Background] Zorad S, Macho L, Jezova D, Fickova M. Partial characterization of insulin resistance in adipose tissue of monosodium glutamate-induced obese rats. Ann N Y Acad Sci. 1997 Sep 20;827:541-5. doi: 10.1111/j.1749-6632.1997.tb51867.x. No abstract available. PMID 9329787
- [Background] Arenas IA, Xu Y, Lopez-Jaramillo P, Davidge ST. Angiotensin II-induced MMP-2 release from endothelial cells is mediated by TNF-alpha. Am J Physiol Cell Physiol. 2004 Apr;286(4):C779-84. doi: 10.1152/ajpcell.00398.2003. Epub 2003 Nov 26. PMID 14644777
- [Background] Benson SC, Pershadsingh HA, Ho CI, Chittiboyina A, Desai P, Pravenec M, Qi N, Wang J, Avery MA, Kurtz TW. Identification of telmisartan as a unique angiotensin II receptor antagonist with selective PPARgamma-modulating activity. Hypertension. 2004 May;43(5):993-1002. doi: 10.1161/01.HYP.0000123072.34629.57. Epub 2004 Mar 8. PMID 15007034
- [Background] Boustany CM, Bharadwaj K, Daugherty A, Brown DR, Randall DC, Cassis LA. Activation of the systemic and adipose renin-angiotensin system in rats with diet-induced obesity and hypertension. Am J Physiol Regul Integr Comp Physiol. 2004 Oct;287(4):R943-9. doi: 10.1152/ajpregu.00265.2004. Epub 2004 Jun 10. PMID 15191907
- [Background] Dal Ponte DB, Fogt DL, Jacob S, Henriksen EJ. Interactions of captopril and verapamil on glucose tolerance and insulin action in an animal model of insulin resistance. Metabolism. 1998 Aug;47(8):982-7. doi: 10.1016/s0026-0495(98)90355-9. PMID 9711996
- [Background] De Mattia G, Ferri C, Laurenti O, Cassone-Faldetta M, Piccoli A, Santucci A. Circulating catecholamines and metabolic effects of captopril in NIDDM patients. Diabetes Care. 1996 Mar;19(3):226-30. doi: 10.2337/diacare.19.3.226. PMID 8742566
- [Background] Engeli S, Gorzelniak K, Kreutz R, Runkel N, Distler A, Sharma AM. Co-expression of renin-angiotensin system genes in human adipose tissue. J Hypertens. 1999 Apr;17(4):555-60. doi: 10.1097/00004872-199917040-00014. PMID 10404958
- [Background] Engeli S, Schling P, Gorzelniak K, Boschmann M, Janke J, Ailhaud G, Teboul M, Massiera F, Sharma AM. The adipose-tissue renin-angiotensin-aldosterone system: role in the metabolic syndrome? Int J Biochem Cell Biol. 2003 Jun;35(6):807-25. doi: 10.1016/s1357-2725(02)00311-4. PMID 12676168
- [Background] Ernsberger P, Koletsky RJ. Metabolic actions of angiotensin receptor antagonists: PPAR-gamma agonist actions or a class effect? Curr Opin Pharmacol. 2007 Apr;7(2):140-5. doi: 10.1016/j.coph.2006.11.008. Epub 2007 Feb 15. PMID 17303473
- [Background] Ferrario CM, Jessup J, Gallagher PE, Averill DB, Brosnihan KB, Ann Tallant E, Smith RD, Chappell MC. Effects of renin-angiotensin system blockade on renal angiotensin-(1-7) forming enzymes and receptors. Kidney Int. 2005 Nov;68(5):2189-96. doi: 10.1111/j.1523-1755.2005.00675.x. PMID 16221218
- [Background] Furuhashi M, Ura N, Higashiura K, Murakami H, Tanaka M, Moniwa N, Yoshida D, Shimamoto K. Blockade of the renin-angiotensin system increases adiponectin concentrations in patients with essential hypertension. Hypertension. 2003 Jul;42(1):76-81. doi: 10.1161/01.HYP.0000078490.59735.6E. Epub 2003 Jun 9. PMID 12796280
- [Background] Goossens GH, Blaak EE, van Baak MA. Possible involvement of the adipose tissue renin-angiotensin system in the pathophysiology of obesity and obesity-related disorders. Obes Rev. 2003 Feb;4(1):43-55. doi: 10.1046/j.1467-789x.2003.00091.x. PMID 12608526
- [Background] Gorzelniak K, Engeli S, Janke J, Luft FC, Sharma AM. Hormonal regulation of the human adipose-tissue renin-angiotensin system: relationship to obesity and hypertension. J Hypertens. 2002 May;20(5):965-73. doi: 10.1097/00004872-200205000-00032. PMID 12011658
- [Background] Guerre-Millo M. Adipose tissue and adipokines: for better or worse. Diabetes Metab. 2004 Feb;30(1):13-9. doi: 10.1016/s1262-3636(07)70084-8. PMID 15029093
- [Background] Haenni A, Berglund L, Reneland R, Anderssson PE, Lind L, Lithell H. The alterations in insulin sensitivity during angiotensin converting enzyme inhibitor treatment are related to changes in the calcium/magnesium balance. Am J Hypertens. 1997 Feb;10(2):145-51. doi: 10.1016/s0895-7061(96)00343-3. PMID 9037321
- [Background] Havel PJ. Update on adipocyte hormones: regulation of energy balance and carbohydrate/lipid metabolism. Diabetes. 2004 Feb;53 Suppl 1:S143-51. doi: 10.2337/diabetes.53.2007.s143. PMID 14749280
- [Background] Henriksen EJ, Jacob S. Modulation of metabolic control by angiotensin converting enzyme (ACE) inhibition. J Cell Physiol. 2003 Jul;196(1):171-9. doi: 10.1002/jcp.10294. PMID 12767053
- [Background] Hotamisligil GS, Shargill NS, Spiegelman BM. Adipose expression of tumor necrosis factor-alpha: direct role in obesity-linked insulin resistance. Science. 1993 Jan 1;259(5091):87-91. doi: 10.1126/science.7678183.
- [Background] Iwai M, Chen R, Imura Y, Horiuchi M. TAK-536, a new AT1 receptor blocker, improves glucose intolerance and adipocyte differentiation. Am J Hypertens. 2007 May;20(5):579-86. doi: 10.1016/j.amjhyper.2006.12.010. PMID 17485025
- [Background] Janke J, Engeli S, Gorzelniak K, Luft FC, Sharma AM. Mature adipocytes inhibit in vitro differentiation of human preadipocytes via angiotensin type 1 receptors. Diabetes. 2002 Jun;51(6):1699-707. doi: 10.2337/diabetes.51.6.1699. PMID 12031955
- [Background] Jankowski V, Vanholder R, van der Giet M, Tolle M, Karadogan S, Gobom J, Furkert J, Oksche A, Krause E, Tran TN, Tepel M, Schuchardt M, Schluter H, Wiedon A, Beyermann M, Bader M, Todiras M, Zidek W, Jankowski J. Mass-spectrometric identification of a novel angiotensin peptide in human plasma. Arterioscler Thromb Vasc Biol. 2007 Feb;27(2):297-302. doi: 10.1161/01.ATV.0000253889.09765.5f. Epub 2006 Nov 30. PMID 17138938
- [Background] Kaplan NM. Hypertension and diabetes. J Hum Hypertens. 2002 Mar;16 Suppl 1:S56-60. doi: 10.1038/sj.jhh.1001344. PMID 11986896
- [Background] Karlsson C, Lindell K, Ottosson M, Sjostrom L, Carlsson B, Carlsson LM. Human adipose tissue expresses angiotensinogen and enzymes required for its conversion to angiotensin II. J Clin Endocrinol Metab. 1998 Nov;83(11):3925-9. doi: 10.1210/jcem.83.11.5276. PMID 9814470
- [Background] Keidar S, Kaplan M, Gamliel-Lazarovich A. ACE2 of the heart: From angiotensin I to angiotensin (1-7). Cardiovasc Res. 2007 Feb 1;73(3):463-9. doi: 10.1016/j.cardiores.2006.09.006. Epub 2006 Sep 19. PMID 17049503
- [Background] Kim S, Iwao H. Molecular and cellular mechanisms of angiotensin II-mediated cardiovascular and renal diseases. Pharmacol Rev. 2000 Mar;52(1):11-34. PMID 10699153
- [Background] Kim S, Moustaid-Moussa N. Secretory, endocrine and autocrine/paracrine function of the adipocyte. J Nutr. 2000 Dec;130(12):3110S-3115S. doi: 10.1093/jn/130.12.3110S. PMID 11110881
- [Background] Mori Y, Itoh Y, Tajima N. Angiotensin II receptor blockers downsize adipocytes in spontaneously type 2 diabetic rats with visceral fat obesity. Am J Hypertens. 2007 Apr;20(4):431-6. doi: 10.1016/j.amjhyper.2006.09.016. PMID 17386352
- [Background] Noshiro T, Way D, McGrath BP. Effect of angiotensin-converting enzyme inhibition on renal norepinephrine spillover rate and baroreflex responses in conscious rabbits. Clin Exp Pharmacol Physiol. 1991 May;18(5):375-8. doi: 10.1111/j.1440-1681.1991.tb01467.x. PMID 1648463
- [Background] Oksa A, Gajdos M, Fedelesova V, Spustova V, Dzurik R. Effects of angiotensin-converting enzyme inhibitors on glucose and lipid metabolism in essential hypertension. J Cardiovasc Pharmacol. 1994 Jan;23(1):79-86. doi: 10.1097/00005344-199401000-00010. PMID 7511740
- [Background] Pinterova L, Krizanova O, Zorad S. Rat epididymal fat tissue express all components of the renin-angiotensin system. Gen Physiol Biophys. 2000 Sep;19(3):329-34. PMID 11316063
- [Background] Pinterova L, Zelezna B, Fickova M, Macho L, Krizanova O, Jezova D, Zorad S. Elevated AT1 receptor protein but lower angiotensin II-binding in adipose tissue of rats with monosodium glutamate-induced obesity. Horm Metab Res. 2001 Dec;33(12):708-12. doi: 10.1055/s-2001-19132. PMID 11753755
- [Background] Rieusset J, Touri F, Michalik L, Escher P, Desvergne B, Niesor E, Wahli W. A new selective peroxisome proliferator-activated receptor gamma antagonist with antiobesity and antidiabetic activity. Mol Endocrinol. 2002 Nov;16(11):2628-44. doi: 10.1210/me.2002-0036. PMID 12403851